CLINICAL TRIAL: NCT01909167
Title: A Randomized Controlled Trial of Internet Based Cognitive Behavioural Therapy (CBT) Versus Treatment as Usual (TAU) for Pregnant Women With Symptoms of Depression
Brief Title: Keeping Well:Online Cognitive Behavioral Therapy (CBT) for Pregnant Women With Depressive Symptoms
Acronym: OnCBTDep
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: CI had other commitments
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13IC0475
Record Dates: First submitted 2013-07-02; First posted 2013-07-26 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Anxiety; Mental Disorders; Postpartum Depression; Depressive Symptoms
Keywords: Pregnancy; symptoms of depression; anxiety; online CBT therapy; treatment as usual; maternal bonding; postnatal period
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders; Depression, Postpartum; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (Active Comparator): Patients randomized to the treatment as usual arm will follow advice by their GP(general practitioner), mental health midwife or perinatal psychiatric team concerning treatment.
  Interventions: Other: Treatment as usual
- Online Cognitive Behavioral Therapy (Active Comparator): CBT treatment: Patients randomized to the online treatment will have, in total, 10 real time individual sessions of 40min each, starting at the 20-23rd gestational week and lasting until 6 weeks postpartum. The therapy will be delivered every two weeks, with a break from the 36th gestational week until the 4th week postpartum.
  Interventions: Behavioral: Online Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Online Cognitive Behavioral Therapy (CBT) — CBT treatment: Patients randomized to the online treatment will have, in total, 10 real time individual sessions of 40min each, starting at the 20-23rd gestational week and lasting until 6 weeks postpartum. The therapy will be delivered every two weeks, with a break from the 36th gestational week until the 4th week postpartum.
  Arms: Online Cognitive Behavioral Therapy
Other: Treatment as usual — Patients randomized to the treatment as usual arm will be advised by their GP,perinatal psychiatric team or mental health midwife concerning treatment.
  Arms: Treatment as usual (TAU)

SUMMARY:
Most depression during pregnancy is undetected and untreated although it is known to be harmful both to the woman herself and her future child. When these mental disorders are detected, psychotherapies remain difficult to access, especially in primary care, despite being effective.Also, prenatal depression is known to be a strong risk factor for postnatal depression and may prejudice the mother-infant relationship. This leads us to the following question: Will individual Cognitive Behavioral Therapy (CBT) delivered online be a more effective treatment for symptoms of depression in pregnant women, than treatment as usual (TAU)?

The proposed randomized controlled trial aims at evaluating the efficacy of internet based cognitive behavioural therapy(CBT) delivered individually via "skype", using video and audio resources, by a fully trained psychotherapist, compared to treatment as usual, in women suffering from symptoms of depression in pregnancy.

Hypothesis The internet based interventions will be more effective at reducing symptoms of depression in pregnant women than treatment as usual, in terms of rates of diagnoses and levels of self rated symptoms of depression.

DETAILED DESCRIPTION:
In the last hundred years there has been a great improvement in the physical care of pregnant women, with a corresponding decline in morbidity and mortality for both mother and child. This same is not true of their psychological and psychiatric care in pregnancy, and this is arguably one of the most important unmet aspects of current obstetrics. Previous research has shown that if a mother has high levels of depression or anxiety during pregnancy, including in later gestation,her child is at about double the risk for ADHD(attention deficit hyperactivity disorder), conduct disorder and emotional problems later in development, as well as increased risk for cognitive delay. Prenatal stress, depression and anxiety contribute an estimated 10-15% of the variance in these outcomes. High levels of antenatal anxiety and depression are frequently co-morbid and have been shown to increase risk for preterm delivery, low birth weight, as well as being a major risk factor for postpartum depression and recurrent maternal depression. This in turn, is also associated with increased risk of long-term emotional and behavioral problems in children.

Over 80% of pregnant women with depression are currently undiagnosed and untreated. Most women prefer non pharmacological treatments during gestation and NICE(National Institute for Health and Care Excellence) clinical guidelines recommend Cognitive Behavioral Therapy (CBT) for the treatment of these disorders at this time. CBT has been shown to be effective for the treatment of depression in general; however there have been no randomized controlled trials with pregnant women. Since they may respond differently, they need to be studied directly. The most cost effective way of delivering personalized CBT is internet based and it can be offered online, individually and in real time. Computerized CBT programs have been developed to improve accessibility, but are inflexible, difficult to adapt to patient's specific needs and are associated to low rates of adherence. So, due to the real need of more accessible psychological therapies in primary care, it is crucial to investigate the efficacy of relatively low cost therapeutic tools to improve and broaden individual patient care in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* To be pregnant
* Less than 20 weeks gestation,
* To have symptoms of depression (EPDS between 12-22),
* To be computer literate,
* To have an online computer at home,
* English speaking and writing,
* Not being in psychiatric or psychological treatment,
* Not having a twin pregnancy,
* Not having undertaken an IVF (In vitro fertilization) procedure,
* Not having the psychiatric problems (based on the patient's notes): psychosis, addiction, history of bipolar disorder, suicidality and other psychiatric diagnoses that do not fall into the affective disorders and/or anxiety disorders spectrum.

Exclusion Criteria:

* Not pregnant
* Having severe symptoms of depression (EPDS above 22),
* Computer illiteracy,
* No access to the internet,
* Not speaking or reading English,
* Already being in psychiatric or psychological treatment,
* Twin pregnancy,
* Having a medical disorder of pregnancy (including abnormal foetus),
* Having undertaken an IVF (In vitro fertilization) procedure,
* Psychiatric factors based on patient's notes: psychosis, addiction, history of bipolar disorder, suicidality and other psychiatric diagnoses that do not fall into the affective disorders and/or anxiety disorders spectrum.
* After birth for baby data: baby born below 35 weeks, baby with any severe disorders. Mothers will continue to be treated if they want to.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Edinburgh Postnatal Depression Scale (EPDS)scores from 20 weeks antenatal to 10 weeks postnatal | Prenatal: 20, 28, 36weeks.Postnatal: 4 and 10 weeks
  The primary outcome will be the change in the EPDS scores from before to after intervention in the Cognitive Behavioral Therapy(CBT) online group compared with treatment as usual (TAU) conditions.

SECONDARY OUTCOMES:
Compliance and dropout rates from 20 weeks antenatal to 4 weeks postnatal | Prenatal: 20, 28, 36 weeks.Postnatal: 4 and 10 weeks
  Secondary outcome will be to assess the compliance and drop out rates in the CBT and TAU group
Changes in anxiety scores from 20 weeks antenatal to 10 weeks postnatal | Prenatal: 20, 28, 36 weeks.Postnatal: 4 and 10 weeks
  Secondary outcome will be the changes in anxiety scores in the CBT and TAU group
Changes in bonding scores at 10 weeks postnatal | Postnatal: 10 weeks
  Secondary outcome will to check the differences in the bonding scores in the CBT and TAU group

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kammerer, PhD, Principal Investigator — Imperial College London
Locations (1):
- Queen Charlotte's and Chelsea Hospital, London, United Kingdom

REFERENCES:
- [Background] Christensen H, Griffiths KM, Mackinnon AJ, Brittliffe K. Online randomized controlled trial of brief and full cognitive behaviour therapy for depression. Psychol Med. 2006 Dec;36(12):1737-46. doi: 10.1017/S0033291706008695. Epub 2006 Aug 29. PMID 16938144
- [Background] Goodman JH. Women's attitudes, preferences, and perceived barriers to treatment for perinatal depression. Birth. 2009 Mar;36(1):60-9. doi: 10.1111/j.1523-536X.2008.00296.x. PMID 19278385
- [Background] Hedegaard M, Henriksen TB, Sabroe S, Secher NJ. Psychological distress in pregnancy and preterm delivery. BMJ. 1993 Jul 24;307(6898):234-9. doi: 10.1136/bmj.307.6898.234. PMID 8369684
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Kessler D, Lewis G, Kaur S, Wiles N, King M, Weich S, Sharp DJ, Araya R, Hollinghurst S, Peters TJ. Therapist-delivered Internet psychotherapy for depression in primary care: a randomised controlled trial. Lancet. 2009 Aug 22;374(9690):628-34. doi: 10.1016/S0140-6736(09)61257-5. PMID 19700005
- [Background] McClure EM, Goldenberg RL, Bann CM. Maternal mortality, stillbirth and measures of obstetric care in developing and developed countries. Int J Gynaecol Obstet. 2007 Feb;96(2):139-46. doi: 10.1016/j.ijgo.2006.10.010. Epub 2007 Feb 1. PMID 17274999
- [Background] National Institute for Clinical Health Excellence (NICE) (2008). Technology appraisal 97: Computerized cognitive behavioural therapy for depression and anxiety (Review of technology appraisal 51), NICE, London.
- [Background] Oates MR. Adverse effects of maternal antenatal anxiety on children: causal effect or developmental continuum? Br J Psychiatry. 2002 Jun;180:478-9. doi: 10.1192/bjp.180.6.478. No abstract available. PMID 12042222
- [Background] O'Connor TG, Heron J, Golding J, Beveridge M, Glover V. Maternal antenatal anxiety and children's behavioural/emotional problems at 4 years. Report from the Avon Longitudinal Study of Parents and Children. Br J Psychiatry. 2002 Jun;180:502-8. doi: 10.1192/bjp.180.6.502. PMID 12042228
- [Background] Talge NM, Neal C, Glover V; Early Stress, Translational Research and Prevention Science Network: Fetal and Neonatal Experience on Child and Adolescent Mental Health. Antenatal maternal stress and long-term effects on child neurodevelopment: how and why? J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):245-61. doi: 10.1111/j.1469-7610.2006.01714.x. PMID 17355398
- [Background] Vesga-Lopez O, Blanco C, Keyes K, Olfson M, Grant BF, Hasin DS. Psychiatric disorders in pregnant and postpartum women in the United States. Arch Gen Psychiatry. 2008 Jul;65(7):805-15. doi: 10.1001/archpsyc.65.7.805. PMID 18606953